CLINICAL TRIAL: NCT00766740
Title: Individual-Patient-Data Pooled-Analysis Comparing Long Term Clinical Outcome in Patients With ST-Elevation Myocardial Infarction Treated With Percutaneous Coronary Intervention With or Without Prior Thrombectomy
Brief Title: Long Term Clinical Efficacy of Thrombectomy Devices in Acute ST Elevation Myocardial Infarction
Acronym: ATTEMPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Francesco Burzotta, MD, PhD, Catholic University of Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSC-001
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Acute Myocardial Infarction
Keywords: ST elevation myocardial infarction; thrombectomy; primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): thrombectomy
  Interventions: Device: thrombectomy devices
- 2 (Active Comparator): Standard PCI
  Interventions: Device: angioplasty

INTERVENTIONS:
Device: thrombectomy devices — mechanical or manual devices able to remove thrombus from the coronary arteries.
  Other Names: DIVER CE; PRONTO; EXPORT; X-SIZER; TVAC; RESCUE; ANGIO-JET
  Arms: 1
Device: angioplasty — percutaneous coronary angioplasty with use of balloon catheters and bare metal stents or drug eluting stents.
  Arms: 2

SUMMARY:
Available data from randomized trials on thrombectomy in patients with ST-elevation myocardial infarction have shown favourable trends on myocardial reperfusion. Better myocardial reperfusion may translate in better late clinical outcome. However, only few data are available on the impact of thrombectomy on long term clinical outcome.

Thus, the investigators designed a collaborative individual patient-data pooled-analysis aimed to assess the long-term clinical outcome in STEMI patients randomized to percutaneous coronary intervention with or without thrombectomy.

DETAILED DESCRIPTION:
Background: Available data from randomized trials on thrombectomy in patients with ST-elevation myocardial infarction have shown favourable trends on myocardial reperfusion. However, only few data are available on the impact of thrombectomy on long term clinical outcome.The first trials on thrombectomy had a too small sample size and a too short follow-up to reliably assess the presence of a clinical benefit.

Only one, recently published, monocentric, randomized trial conducted on 1071 patients with STEMI, the TAPAS study, showed an advantage of thrombus-aspiration use in terms of mortality at one year follow-up.

To extend the investigation on this issue to a larger population, we have designed a pooled analysis of the individual patient data of prospective randomized trials comparing standard PCI with or without thrombectomy to evaluate the impact of thrombectomy use on long term clinical outcome.

Methods: After a thorough database search, all 15 principal investigators of 17 randomized trials comparing thrombectomy with standard PCI in patients with STEMI were contacted. All 10 principal investigators authoring 11 randomized trials who agreed to participate the study have been asked to complete a structured database including a series of key baseline clinical and angiographic data (sex, age, diabetes, rescue PCI, usage of IIb/IIIa-inhibitors, infarct related artery (LAD or LCX or RCA), multivessel disease, base-line TIMI flow 0 or 1 (yes or no), time from symptoms to balloon/cath-lab, thrombectomy device used (name of the device, for example Export catheter),device efficacy (device able to reach and treat the culprit lesion)) and also to update the clinical follow-up of each patient enrolled in the corresponding trial at one year or more.

Actually we have closed the data collection and we have the requested data with the updated clinical follow-up data of 11 randomized studies (REMEDIA trial, PIHRATE trial, X-AMINE ST trial, De Luca et al. trial, Noel et al. trial, EXPIRA trial, VAMPIRE trial, TAPAS trial, Kaltoft et al. trial, DEAR-MI trial, Antoniucci et al. trial).

The primary end point of this pooled analysis is the comparison of survival between patients randomized to PCI with thrombectomy or PCI without thrombectomy. The secondary end-points are survival free from myocardial infarction (MI), target lesion revascularization (TLR), major adverse coronary events (MACE: death + MI + TLR) and death + MI between patients randomized to PCI with thrombectomy or PCI without thrombectomy.

A pre-defined subgroup analysis is planned considering the following variables: diabetes, rescue PCI, IIb/IIIa-inhibitors use, time-to-reperfusion, infarct related artery, pre-PCI TIMI flow and type of thrombectomy device used.

Implications: This study will be able to provide useful data about the impact of the reported improved myocardial perfusion associated with thrombectomy on the long-term clinical outcome in patients with STEMI.

ELIGIBILITY:
Inclusion criteria for selected studies who entered this pooled analysis were:

* Comparison of PCI with Thrombectomy with Standard PCI in patients with STEMI
* Randomized treatment allocation

Exclusion criteria was:

* Equivocal treatment allocation process

About the clinical and angiographic inclusion and exclusion criteria they were different for each single randomized trial that entered this pooled analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2686 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
All cause mortality | one year

SECONDARY OUTCOMES:
Major adverse coronary events (MACE: death + MI (myocardial infarction) + TLR (target lesion revascularization) | one year
Myocardial infarction | one year
Death + myocardial infarction | one year

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, MD, PhD, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Vlaar PJ, Svilaas T, van der Horst IC, Diercks GF, Fokkema ML, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Cardiac death and reinfarction after 1 year in the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS): a 1-year follow-up study. Lancet 2008; 371(9628):1915-20. Antoniucci D, Valenti R, Migliorini A, Parodi G, Memisha G, Santoro GM, Sciagra R. Comparison of rheolitic thrombectomy before direct infarct artery stenting versus direct stenting alone in patients undergoing percutaneous coronary intervention of acute myocardial infarction. Am J Cardiol 2004,93:1033-35. Dudek D, Mielecki W, Legutko J, Chyrchel M, Sorysz D, Bartus S, Rzeszutko L, Dubiel JS. Percutaneous thrombectomy with the RESCUE system in acute myocardial infartion. Kardiol Pol 2004;61:523-33. Burzotta F, Trani C, Romagnoli E, Mazzari MA, Rebuzzi AG, De Vita M, Garramone B, Giannico F, Niccoli G, Biondi-Zoccai GG, Schiavoni G, Mongiardo R, Crea F. Manual thrombus-aspiration improves myocardial reperfusion: the randomized evaluation of the effect of mechanical reduction of distal embolization by thrombus-aspiration in primary and rescue angioplasty (REMEDIA) trial. J Am Coll Cardiol. 2005 ;46(2):371-6. Lefevre T, Garcia E, Reimers B, Lang I, di Mario C, Colombo A, Neumann FJ, Chavarri MV, Brunel P, Grube E, Thomas M, Glatt B, Ludwig J; X AMINE ST Investigators. X-sizer for thrombectomy in acute myocardial infarction improves ST-segment resolution: results of the X-sizer in AMI for negligible embolization and optimal ST resolution (X AMINE ST) trial. J Am Coll Cardiol 2005;46:246-52. Noel B, Morice MC, Lefevre T et al. Thrombus aspiration in acute ST-elevation myocardial infarction: a randomized controlled trial. Circulation 2005; 112 (Suppl. II): 519. Silva-Orrego P, Colombo P, Bigi R, Gregori D, Delgado A, Salvade P, Oreglia J, Orrico P, de Biase A, Piccalò G, Bossi I, Klugmann S. Thrombus aspiration before primary angioplasty improves myocardial reperfusion in acute myocardial infarction: the DEAR-MI (Dethrombosis to Enhance Acute Reperfusion in Myocardial Infarction) study. J Am Coll Cardiol 2006 17;48:1552-9. Ikari Y, Kawano S, Sakurada M, et al. Thrombus aspiration prior to coronary intervention improves myocardial microcirculation in patients with ST elevation acute myocardial infarction, the VAMPIRE Study. Circulation 2005;112 [Suppl., abstr]. Kaltoft A, Bottcher M, Nielsen SS, Hansen HH, Terkelsen C, Maeng M, Kristensen J, Thuesen L, Krusell LR, Kristensen SD, Andersen HR, Lassen JF, Rasmussen K, Rehling M, Nielsen TT, Botker HE. Routine thrombectomy in percutaneous coronary intervention for acute ST-segment-elevation myocardial infarction: a randomized, controlled trial. Circulation 2006;114:40-7. De Luca L, Sardella G, Davidson CJ, De Persio G, Beraldi M, Tommasone T, Mancone M,Nguyen BL, Agati L, Gheorghiade M, Fedele F. Impact of intracoronary aspiration thrombectomy during primary angioplasty on left ventricular remodelling in patients with anterior ST elevation myocardial infarction. Heart 2006;92:951-7. Svilaas T, Vlaar PJ, van der Horst IC et al. Thrombus Aspiration during Primary Percutaneous Coronary Intervention. N Engl J Med 2008;358: 557-67. Dudek D et al. Polish-Italian-Hungarian Randomized ThrombEctomy Trial. PHIRATE trial; Expert slide presentation from Late Breaking Clinical Trials, TCT 2007. Sardella G et al. Impact of thrombectomy with EXPort catheter in Infarct Related Artery on procedural and clinical outcome in patients with AMI. (EXPIRA Trial); Expert slide presentation from Late Breaking Clinical Trials, TCT 2007. Chevalier B. Export Study; Expert slide presentation from Late Breaking Clinical Trials, TCT 2007.
- [Derived] Burzotta F, De Vita M, Gu YL, Isshiki T, Lefevre T, Kaltoft A, Dudek D, Sardella G, Orrego PS, Antoniucci D, De Luca L, Biondi-Zoccai GG, Crea F, Zijlstra F. Clinical impact of thrombectomy in acute ST-elevation myocardial infarction: an individual patient-data pooled analysis of 11 trials. Eur Heart J. 2009 Sep;30(18):2193-203. doi: 10.1093/eurheartj/ehp348. Epub 2009 Sep 2. PMID 19726437